CLINICAL TRIAL: NCT01978977
Title: Maintenance Bevacizumab or Observation After Taxane Based First Line Chemotherapy Plus Bevacizumab in Women With HER2-Negative Metastatic Breast Cancer. An Observational Study.
Brief Title: Maintenance Bevacizumab or Observation After Taxane Based First Line Chemotherapy In Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: CT/10.17
Record Dates: First submitted 2013-11-03; First posted 2013-11-08 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Metastatic Breast Cancer
Keywords: mBC; HER2 negative; Chemotherapy; Anti-angiogenic agent; Bevacizumab; 1st Line
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Avastin regimens: Patients who are going to receive chemotherapy plus Avastin (bevacizumab)

SUMMARY:
Investigators propose to assess,the safety and tolerability profile (number of participants with adverse events)of bevacizumab (Avastin) when combined with standard chemotherapy as first line treatment of patients with metastatic Breast Cancer.

DETAILED DESCRIPTION:
Nowadays in clinical practice patients with previously untreated metastatic breast cancer often receive taxane-based chemotherapy (paclitaxel or docetaxel) in combination with bevacizumab as it has been shown to increase progression-free survival. There is currently minimal information whether bevacizumab should be given as maintenance therapy after discontinuation of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥18 years
* Patients with histologically or cytologically confirmed, HER2-negative, metastatic Breast Cancer
* No prior first line treatment for metastatic Breast Cancer
* Previous hormonotherapy for metastatic Breast Cancer is allowed
* One or more measurable lesions (≥1cm in diameter with spiral CT scan or ≥2cm with conventional techniques) according to RECIST criteria
* ECOG performance status ≤2
* Adequate haematological, renal and hepatic function
* Urine protein <2+ (dipstick)
* Life expectancy of ≥12 weeks

Exclusion Criteria:

* Previous first line treatment for metastatic colorectal cancer(progression >12 months after the end of adjuvant treatment)
* Previous radiotherapy to target lesions
* Patients with brain metastases and/or cancerous meningitis
* Presence or history of other neoplasm except properly treated basal cell skin cancer or in situ cervical carcinoma
* Patients participating in interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinics for cancer prevention
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2011-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Every 2 or 3 weeks up to 12 or 18 weeks
  In this observational study investigators are going to assess standard schedules in which administration was every 2 or 3 weeks

SECONDARY OUTCOMES:
Number of Participants with Response Rate | Disease evaluation at Week 3 or at week 6
  In this observational study investigators are going to assess standard schedules in which the disease evaluation was performed every 3 or 6 weeks
Percentage of Patients with Progression Free Survival | 1 year
Patients Overall Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Georgoulias, MD, Principal Investigator — Hellenic Oncology Research Group
Locations (6):
- Greece (6):
  - University Hospital of Crete, Dep of Medical Oncology, Heraklion, Crete
  - University General Hospital of Alexandroupolis, Dept. of Medical Oncology, Alexandroupoli
  - "IASO" General Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens, Athens
  - "Metaxa's" Anticancer Hospital of Piraeus, 1st Dep of Medical Oncology, Piraeus
  - "Theagenion" Anticancer Hospital of Thessaloniki, 2nd Dep of Medical Oncology, Thessaloniki